CLINICAL TRIAL: NCT05313672
Title: Inspiratory Effort and Respiratory Mechanics in Spontaneously Breathing Patients With Acute Exacerbation of Idiopathic Pulmonary Fibrosis: a Matched Control Study
Acronym: IERATIC
Status: Active, not recruiting | Type: Observational
Sponsor: Roberto Tonelli (Other)
Responsible Party: Sponsor-Investigator, Roberto Tonelli, Principal investigator, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Other Study IDs: UModenaReggio21
Record Dates: First submitted 2022-03-28; First posted 2022-04-06 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Inspiratory effort; Esophageal manometry; Non-invasive mechanical ventilation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IPF patients with UIP pattern requiring NIV
- ARDS patients requiring NIV

SUMMARY:
Idiopathic pulmonary fibrosis is a life-threatening lung disease characterized by progressive deterioration of lung function and a median survival time of 3-5 years from diagnosis. The onset of an acute deterioration (AE) of respiratory function, the so called acute exacerbation of IPF (AE-IPF), may lead to severe hypoxemia, further worsening prognosis. During these events, the typical usual interstitial pneumonia pattern (UIP) - the radiologic and histologic hallmark of IPF- is overlapped with diffuse alveolar damage (DAD), sharing similarities with the acute respiratory distress syndrome (ARDS) and often requiring respiratory assistance. Several studies show that the need for mechanical ventilation (MV) is associated with high mortality in IPF patients, probably due to the pathophysiological properties of UIP-like fibrotic lung (i.e. collapse induration areas, elevated lung elastance, high inhomogeneity) that make it more susceptible to ventilatory-induced lung injury (VILI). It has been theorized that the application of PEEP on a UIP-like lung pattern can determine the protrusion of the most distensible areas through a dense anelastic fibrotic tissue circles, causing increased rigidity, worsening compliance, and thus enabling tissue breakdown. In this scenario, non-invasive mechanical ventilation (NIV) may therefore represent an alternative option to assist these patients, although no specific recommendations have been made so far. In patients with ARDS, the efficacy of NIV in reducing the patient's inspiratory effort early after its application has been related to a favorable clinical outcome. Indeed, the mitigation of respiratory drive might have resulted in a lower risk for the self-inflicted lung injury (SILI) during spontaneous breathing, whose onset is very likely to worse outcomes of patients undergoing acute respiratory failure (ARF).

To date no data available on the inspiratory effort and the lung mechanics in patients with AE-IPF either during unassisted of assisted spontaneous breathing. Aim of this study was then to compare respiratory mechanics, at baseline and 2-h following NIV application, in AE-IPF and ARDS patients matched for severity.

ELIGIBILITY:
Inclusion Criteria:

previously established diagnosis of IPF; occurring acute exacerbation of IPF as defined by an acute, clinically significant respiratory deterioration characterized by evidence of new widespread alveolar abnormality on chest CT scan (12); age >18 years; presence of ARF with PaO2/FiO2 ratio <200 mmHg despite HFNC (set with at least 60 L/min and FiO2 higher than 0.6); suitability for a NIV trial according to the attending staff; consent to measure esophageal pressure.

Exclusion Criteria:

* acute cardiogenic pulmonary edema,
* concomitant hypercapnic respiratory failure (PaCO2 >45 mmHg) of any etiology,
* neuromuscular disease or chest wall deformities,
* home long-term oxygen therapy,
* intolerance or contraindication to NIV, such as the need for immediate endotracheal intubation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with IPF developing AE consecutively admitted to the Respiratory Intensive Care Unit and the Intensive Care Unit of the University Hospital of Modena over the period August 1st, 2016 to January 1th, 2022 were prospectively considered eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Inspiratory effort in IPF patients | On respiratory intensive care unit admission
  Assessment of esophageal pressure swing in IPF patients during acute exacerbation of disease as compared to ARDS

SECONDARY OUTCOMES:
Respiratory mechanics change after NIV application in IPF patients acute exacerbation | 2 hours
  Respiratory mechanics change after NIV application in IPF patients acute exacerbation as compared to ARDS

IPD SHARING:
Plan to Share IPD: Undecided